CLINICAL TRIAL: NCT05638386
Title: Effect of Plugging the Registration Pin Tract in Robotic-assisted Knee Surgery
Status: Completed | Type: Observational
Sponsor: Reinier Haga Orthopedisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: OC-2022-002
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-11

CONDITIONS: Arthropathy of Knee; Complication of Surgical Procedure
Keywords: Robotic-assisted surgery; Bone plug

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who underwent a robotic-assisted total knee arthroplasty with the use of bone plugs
  Interventions: Procedure: Bone plug
- Patients who underwent a robotic-assisted total knee arthroplasty without the use of bone plugs

INTERVENTIONS:
Procedure: Bone plug — The investigational treatment is the use of a bone plug in the two drill-holes in the tibia, made by two pins for securing the tibial array to the bone. The pins that are used for this, are 4.0mm wide. The bone plug that is used to fill the drill-holes of tibia, is obtained from the bone that is removed during the operation to make place for the new prosthesis. A piece as wide as the drill-hole is cut off the recessed bone and put into this hole. After this, the wound is closed using surgical staples.
  Groups: Patients who underwent a robotic-assisted total knee arthroplasty with the use of bone plugs

SUMMARY:
Introduction: Complications of robotic-assisted total knee arthroplasty (TKA) seem to be rare and consist mainly of infections or fractures. In the Reinier Haga Orthopedisch Centrum (RHOC), postoperative bleeding is experienced to be a complication that often occurs, mainly at the tibial wounds of the registration pins used in robotic-assisted TKA. This often results in longer hospital stay and might interfere with the current fast track knee surgery by a delayed discharge. To overcome this complication, nowadays bone plugs are used in the two drill-holes. Currently, it is unknown whether these bone plugs reduces the incidence of postoperative bleeding.

Objective: To evaluate the incidence of postoperative bleeding in patients that underwent a robotic-assisted TKA and received bone plugs in the two drill-holes in the tibia, compared to patients that underwent the same operation but did not receive bone plugs.

Study design: Retrospective, inventory study

Study population: All patients that underwent a robotic-assisted TKA in the RHOC from December 2020 till October 2022.

Intervention: In the past, some patients that underwent a robotic-assisted TKA received a bone plug in the two tibial drill-holes. This bone is collected from the excess bone that is removed during the operation.

Main study parameters/endpoints: Incidence of postoperative bleeding in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Underwent robotic-assisted total knee arthroplasty between December 2020 and October 2022 with or without the use of bone plugs
* Does not object against use of medical data

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent robotic-assisted total knee arthroplasty in the RHOC between December 2020 and October 2022
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Number of patients with postoperative bleeding | December 2020 - October 2022

SECONDARY OUTCOMES:
Length of hospital stay | December 2020 - October 2022
Complications | December 2020 - October 2022
Reasons which might lengthen hospital stay | December 2020 - October 2022

CONTACTS AND LOCATIONS:
Locations (1):
- RHOC, Zoetermeer, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided